CLINICAL TRIAL: NCT06910852
Title: Hepatic and Portal Vein Transection by Vascular Stapler in Open Living Donor Hepatectomy
Status: Completed | Type: Observational
Sponsor: Abdalla Bashir, MD (Other)
Responsible Party: Sponsor-Investigator, Abdalla Bashir, MD, MD, Jordan Hospital
Organization: Jordan Hospital (Other)
Other Study IDs: STAPLER/TXS/11_20
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Vascular stapler — the utilization of vascular staplers for the division of the right portal and hepatic veins in patients undergoing right lobe liver donation for living donor liver transplantation

SUMMARY:
To enhance donor safety in living donor liver transplantation (LDLT), the use of vascular staplers for the division of the right portal and hepatic veins in patients undergoing right lobe liver donation has been introduced. This study examines the application of vascular staplers in LDLT and assesses the subsequent feasibility and safety outcomes for donors.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open living donor hepatectomy
* Age ≥ 18 years, ≤ 80 years
* Written informed consent

Exclusion Criteria:

* None.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open living donor hepatectomy at Jordan Hospital.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Post-operative complications (Clavien-Dindo classification) | From enrollment to the end of treatment at 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan Hospital Amman, Amman, Amman Governorate, Jordan

IPD SHARING:
Plan to Share IPD: No